CLINICAL TRIAL: NCT01658930
Title: A Randomized Phase III Trial Comparing Radical Hysterectomy and Pelvic Node Dissection vs Simple Hysterectomy and Pelvic Node Dissection in Patients With Low-Risk Early Stage Cervical Cancer (SHAPE)
Brief Title: Radical Versus Simple Hysterectomy and Pelvic Node Dissection With Low-risk Early Stage Cervical Cancer
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Gynecologic Cancer Intergroup (GCIG) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Korean Gynecologic Oncology Group (Other); Dutch Gynaecological Oncology Group (Other); Cancer Trials Ireland (Network); Arbeitsgemeinschaft Gynaekologische Onkologie Austria (Other); Belgian Gynaecological Oncology Group (Other); ARCAGY/ GINECO GROUP (Other); Institute of Cancer Research, United Kingdom (Other); Shanghai Cancer Centre (Other); P. Herzen Moscow Oncology Research Institute (Other Government); Arbeitsgemeinschaft Gynaekologische Onkologie Studiengruppe Ovarialkarzinom Germany (Other); Institut Universitaire du Cancer de Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX5
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2024-11-22 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical Hysterectomy (Active Comparator)
  Interventions: Procedure: Radical Hysterectomy + pelvic lymph node dissection
- Simple Hysterectomy (Experimental)
  Interventions: Procedure: Simple hysterectomy + pelvic lymph node dissection

INTERVENTIONS:
Procedure: Radical Hysterectomy + pelvic lymph node dissection — This procedure may be performed abdominally, laparoscopically, robotically or vaginally. The uterus, cervix, medial 1/3 of parametria, 2cm of the uterosacral ligaments and upper 1-2cm of the vagina are to be removed en bloc. The uterine artery is ligated laterally to the ureters and the ureters are unroofed to the ureterovesical junction.
  Arms: Radical Hysterectomy
Procedure: Simple hysterectomy + pelvic lymph node dissection — This procedure may be performed abdominally, laparoscopically, robotically or vaginally. Extrafascial hysterectomy involves removal of the uterus with cervix without adjacent parametria. The uterine arteries are transected medial to the ureters at the level of the isthmus and the uterosacral ligaments are transected at the level of the cervix. Surgeons should pay special attention to make sure that the whole cervix is removed. As such, a maximum of 0.5 cm of vaginal cuff can be removed to ensure the complete removal of the cervix.
  Arms: Simple Hysterectomy

SUMMARY:
The reason this study is being done is to see if a simple hysterectomy is as good as a radical hysterectomy in preventing cancer of the cervix from returning, and whether, because less tissue surrounding the uterus is removed during surgery, there are fewer side-effects after the surgery and in the long-term.

DETAILED DESCRIPTION:
At this time, it is not clear which of these approaches best balances the desire to prevent cancer of the cervix from returning with the risks of side effects after surgery and in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma, squamous, or adenosquamous cancer of the cervix. Diagnosis has been made by LEEP, cone or cervical biopsy and has been reviewed and confirmed by the local reference gynecological pathologist.
* Patient has been classified as low-risk early-stage cervical cancer. These patients include:

  • FIGO Stage IA2 [FIGO Annual Report, 2009], defined as:

  o evidence of disease by microscopy;
* for patients who underwent a LEEP or cone:

  * histologic evidence of depth of stromal invasion > 3.0 and ≤ 5.0 mm based on the local reference pathologist's measurement of the LEEP or cone specimen NB: the maximum depth of stromal invasion must be ≤ 10 mm.
  * histologic evidence of lateral extension that is ≤ 7.0 mm based on the local reference pathologist's measurement of the LEEP or cone specimen; and
  * negative margins (patients with positive margins are considered IB1, see below)
* for patients who underwent a cervical biopsy only:

  * radiologic evidence of less than 50% stromal invasion based on pelvic MRI

    • FIGO Stage IB1 [FIGO Annual Report, 2009] with favorable (low risk) features, defined as:
  * measured stromal invasion and lateral extension that meet the criteria for IA2 (see above) but with positive margins;
  * evidence of disease by clinical exam; lesion must clinically measure ≤ 20 mm
  * evidence of disease by microscopy;
* for patients who underwent a LEEP or cone:

  * histologic evidence of depth of stromal invasion between 5.1-10 mm and/or lateral extension between 7.1-20.0 mm based on the local reference pathologist's measurement of the LEEP or cone specimen
* for patients who underwent a cervical biopsy only:
* radiologic evidence of less than 50% stromal invasion based on pelvic MRI
* lateral extension ≤ 20 mm based on clinical exam or radiologic imaging.

In addition to above criteria on maximal stromal invasion of ≤ 10 mm, the lesion must be no larger than 20 mm in any dimension by any assessment method (MRI, clinical or histological exam). To ensure patients meet this criterion, investigators may need to sum the lesion measurements from biopsy and other methods that evaluate it in the same plane.

Patients are eligible irrespective of the presence or absence of lymph-vascular space involvement (LVSI).

* Physical examination, recto-vaginal examination and visualization of the cervix by speculum or colposcopic examination have been done after the initial diagnostic procedure (LEEP, cone or biopsy) and prior to randomization.
* Chest x-ray or CT scan of chest AND pelvic MRI* done after initial diagnostic procedure (LEEP, cone or biopsy) and prior to randomization.

The CT should be a 16 slice (or higher) helical scanner. Oral and intravenous contrasts are preferred (unless there is a contraindication to the use of contrast) with scan obtained in the portal phase at a slice thickness of 5mm or lower Pelvic MRI should be performed on a 1.5 or 3 Tesla magnet with pelvic phased-array coils. The MR pulse sequences will consist of T1 gradient echo in the axial plane at 5 mm slice thickness and fast spin echo in the axial, sagittal, and coronal planes at 4 mm slice thickness. The short axis (perpendicular to the tumour's long axis) with a 3 mm slice thickness is required in the best plane to show the maximum thickness of stromal invasion. Use of an anti-peristaltic agent is mandatory while intravenous use of gadolinium or diffusion-weighted imaging (DWI) is optional.

* Note: pelvic MRI is optional if the patient has stage IA2 disease and underwent a LEEP or cone.

* After consideration of a patient's medical history, physical examination and laboratory testing, patients must be suitable candidates for surgery as defined by the attending physician / investigator.
* Patients must have no desire to preserve fertility.
* Patients fluent in English or French must be willing to complete the Quality of Life Questionnaire. The baseline assessments must be completed within 6 weeks prior to randomization. Inability (illiteracy in English or French, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible. As additional GCIG groups join the study, more translations of some of the questionnaires may be added.

Patients fluent in English or French who reside in Canada and the United Kingdom must agree to participate in the economic evaluation component of this trial and complete the Health Economics Questionnaire. Similarly, patients fluent in English or French accrued from other GCIG groups who are participating in the economic evaluation must be willing to complete the Health Economics Questionnaires.

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Surgery is to be done within 20 weeks of initial diagnosis (NO EXCEPTIONS). The 20-week period includes time required for diagnosis, referral, diagnostic staging, randomization and scheduling of the surgical procedure.
* Patients must be ≥ 18 years old.

Exclusion Criteria:

* Patients with FIGO 1A1 disease [FIGO Annual Report, 2009].
* History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours, Hodgkin's lymphoma or non-Hodgkin's lymphoma curatively treated with no evidence of disease for > 5 years.
* Patients with evidence of lymph node metastasis on preoperative imaging or histology.
* Patients who have had or will receive neoadjuvant chemotherapy.
* Patients who are pregnant.
* Patients for whom adjuvant radiation and/or chemotherapy is planned.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 700 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2023-03-11 (Actual); Study Completion 2024-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Plante, Study Chair — Canadian Cancer Trials Group; Gwenael Ferron, Study Chair — France-GINECO; Jae-Weon Kim, Study Chair — Korean Gynecology Oncology Group; Christian Marth, Study Chair — Arbeitsgemeinschaft Gynaekologische Onkologie Austria; John Tidy, Study Chair — Institute of Cancer Research, United Kingdom; Noreen Gleeson, Study Chair — Ireland Co-operative Oncology Research Group; Frederic Goffin, Study Chair — Belgian Gynaecological Oncology Group; Cor de Kroon, Study Chair — The Dutch Gynecological Oncology Group (DGOG); Xiaohua Wu, Study Chair — Fudan University; Sven Mahner, Study Chair — AGO Germany; Brynhildur Eyjolfsdottir, Study Chair — Oslo University Hospital; Alexey Shevchuk, Study Chair — Hertzen Institute, Moscow
Locations (87):
- Austria (7):
  - Barmherzige Brueder Graz, Graz
  - Medical University of Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - LKH Leoben, Leoben
  - Landes- Frauen- und Kinderklinik Linz, Linz
  - LKH Salzburg, Salzburg
  - Medical University of Vienna, Vienna
- Belgium (3):
  - UZ Leuven, Leuven, Vlaams-Brabant
  - CHR de la Citadelle liege, Liège
  - CHU Sart Tilman Liege, Liège
- Canada (16):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Clinical Research Unit at Vancouver Coastal, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - London Regional Cancer Program, London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Greenfield Park, Quebec
  - CIUSSS de l'Est-de-I'lle-de-Montreal, Montreal, Quebec
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Québec, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec
- Shanghai Cancer Center, Shanghai, China
- France (28):
  - CHU Amiens, Amiens
  - Institut Bergonie Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - CHU de Chambery, Chambéry
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Centre Jean Perrin - Clermont-Ferrand, Clermont-Ferrand
  - Centre Georges Francois Leclerc - Dijon, Dijon
  - CHU de Dijon, Dijon
  - Centre Oscar Lambret - Lille, Lille
  - CHRU de Lille, Lille
  - CHU Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - Centre Leon Berard - Lyon, Lyon
  - Institut Paoli Calmettes - Marseille, Marseille
  - Institut Regional du Cancer de Montpellier, Montpellier
  - Institut Arnault Tzank - Mougins, Mougins
  - CHU de Nice, Nice
  - CHU de Nimes, Nîmes
  - Hopital Europeen Georges Pompidou - Paris, Paris
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - Clinique Mutualiste de la Sagesse - Rennes, Rennes
  - Clinique Mathilde - Rouen, Rouen
  - ICO - Rene Gauducheau, Saint-Herblain
  - CHU de Strasbourg, Strasbourg
  - CHU de Bordeaux, Talence
  - Institut Claudius Regaud - Toulouse, Toulouse
  - CHRU de Tours, Tours
- Germany (21):
  - Hochtaunus-Kliniken gGmbH, Bad Homburg
  - DRK Kliniken Berlin Koepenick, Berlin
  - DRK Klinikum Berlin Westend, Berlin
  - Martin-Luther-Krankenhaus Berlin, Berlin
  - GYNAEKOLOGICUM Bremen, Bremen
  - Universitaetsfrauenklinik Duesseldorf, Düsseldorf
  - Kaiserswerther Diakonie - Florence-Nightingale-Krankenhaus, Düsseldorf
  - Kliniken Essen Mitte, Essen
  - Universitaetsfrauenklinik Freiburg, Freiburg im Breisgau
  - Universitaetsfrauenklinik Greifswald, Greifswald
  - Universitaetsklinikum Hamburg - Eppendorf, Hamburg
  - Agaplesion Diakonieklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum des Saarlandes, Homburg-Saar
  - Universitaetsfrauenklinik Jena, Jena
  - Universitaetsfrauenklinik Luebeck, Lübeck
  - Universitaetsfrauenklinik Mainz, Mainz
  - Klinikum der Universitaet Muenchen - LMU Campus Grosshadern, München
  - Universitaetsfrauenklinik Tuebingen, Tübingen
  - Universitaetsfrauenklinik Ulm, Ulm
  - Marien-Hospital Witten, Witten
- St James Hospital, Dublin, Leinster, Ireland
- Netherlands (2):
  - LUMC, Leiden
  - Erasmus MC, Rotterdam
- Oslo University Hospital, Oslo, Postboks 4953 Nydalen, Norway
- Hertzen Moscow Scientific Research, Moscow, Russia
- United Kingdom (6):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Southend University Hospital, Westcliff-on-Sea, Essex
  - East Kent Hospitals University NHS Foundation Trust, Canterbury, Ethelbert Road
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, Glossop Road
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough, Marton Road
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Plante M, Kwon JS, Ferguson S, Samouelian V, Ferron G, Maulard A, de Kroon C, Van Driel W, Tidy J, Williamson K, Mahner S, Kommoss S, Goffin F, Tamussino K, Eyjolfsdottir B, Kim JW, Gleeson N, Brotto L, Tu D, Shepherd LE; CX.5 SHAPE investigators; CX.5 SHAPE Investigators. Simple versus Radical Hysterectomy in Women with Low-Risk Cervical Cancer. N Engl J Med. 2024 Feb 29;390(9):819-829. doi: 10.1056/NEJMoa2308900. PMID 38416430
- [Derived] Kwon JS, McTaggart-Cowan H, Ferguson SE, Samouelian V, Lambaudie E, Guyon F, Tidy J, Williamson K, Gleeson N, de Kroon C, van Driel W, Mahner S, Hanker L, Goffin F, Berger R, Eyjolfsdottir B, Kim JW, Brotto LA, Pataky R, Yeung SST, Chan KKW, Cheung MC, Ubi J, Tu D, Shepherd LE, Plante M. Cost-effectiveness analysis of simple hysterectomy compared to radical hysterectomy for early cervical cancer: analysis from the GCIG/CCTG CX.5/SHAPE trial. J Gynecol Oncol. 2024 Nov;35(6):e117. doi: 10.3802/jgo.2024.35.e117. Epub 2024 Oct 18. PMID 39453395
- [Derived] Ferguson SE, Brotto LA, Kwon J, Samouelian V, Ferron G, Maulard A, Kroon C, Driel WV, Tidy J, Williamson K, Mahner S, Kommoss S, Goffin F, Tamussino K, Eyjolfsdottir B, Kim JW, Gleeson N, Tu D, Shepherd L, Plante M. Sexual Health and Quality of Life in Patients With Low-Risk Early-Stage Cervical Cancer: Results From GCIG/CCTG CX.5/SHAPE Trial Comparing Simple Versus Radical Hysterectomy. J Clin Oncol. 2025 Jan 10;43(2):167-179. doi: 10.1200/JCO.24.00440. Epub 2024 Oct 1. PMID 39353164
- [Derived] Boisen M, Guido R. Emerging Treatment Options for Cervical Dysplasia and Early Cervical Cancer. Clin Obstet Gynecol. 2023 Sep 1;66(3):500-515. doi: 10.1097/GRF.0000000000000790. Epub 2023 Jul 25. PMID 37650664

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radical Hysterectomy | Simple Hysterectomy
Started | 350 | 350
Completed | 350 | 350
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomized to this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Radical Hysterectomy | Simple Hysterectomy | Total
Number analyzed (Participants) | 350 | 350 | 700
Age, Continuous [Median (Full Range); unit: years] | 45 [24 to 80] | 42 [26 to 77] | 44 [24 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 350 | 350 | 700
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 19 | 22 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 261 | 264 | 525
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 64 | 59 | 123
Region of Enrollment [Number; unit: participants]
  Canada | 92 | 94 | 186
  Austria | 15 | 13 | 28
  Netherlands | 53 | 57 | 110
  Belgium | 20 | 20 | 40
  Norway | 11 | 9 | 20
  China | 0 | 2 | 2
  Ireland | 7 | 7 | 14
  United Kingdom | 49 | 53 | 102
  France | 64 | 58 | 122
  Germany | 29 | 27 | 56
  Russia | 1 | 1 | 2
  South Korea | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Recurrence Rate at 3 Years
Description: Pelvic recurrence rate at 3 years was estimated by 1-the Kaplan-Meier estimate for the probability of pelvic relapse free survival (PRFS) at 3 years. PRFS was defined as the time from randomization to the time when a recurrence within the pelvic field was first documented. Patients who had a relapse outside of the pelvic field documented or died before the documentation of a pelvic relapse were censored at the time of first documented extra-pelvic relapse or death. The pelvic relapse free survival of patients who were alive without any relapse at the time of final analysis was censored at the last known alive.
Time Frame: 3 years
Population: All patients randomized.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Radical Hysterectomy | Simple Hysterectomy
Number analyzed (Participants) | 350 | 350
percentage of participants | 2.17 [0.84 to 3.50] | 2.52 [1.07 to 3.97]
Statistical Analysis 1: Comparison: Radical Hysterectomy vs Simple Hysterectomy; Test type: Non-Inferiority — Margin of inferiority in the difference of 3 year pelvic recurrence rates between simple and radical hysterectomy group was 4%; Mean Difference (Final Values) = 0.0035, 90% CI 2-sided [-0.0162 to 0.0232] — Difference between simple and radical hysterectomy groups

2. Secondary Outcome: Pelvic Relapse-free Survival
Description: It was defined as the time from randomization to the time when a recurrence within the pelvic field was first documented. Patients who had a relapse outside of the pelvic field documented or died before the documentation of a pelvic relapse were censored at the time of first documented extra-pelvic relapse or death. The pelvic relapse free survival of patients who were alive without any relapse at the time of final analysis was censored at the last known alive. 3 year pelvic relapse-free survival was estimated by Kaplan-Meier method.
Time Frame: 3 years
Population: All patients randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radical Hysterectomy | Simple Hysterectomy
Number analyzed (Participants) | 350 | 350
percentage of participants | 97.5 [95.9 to 99.1] | 97.8 [96.2 to 99.4]
Statistical Analysis 1: Comparison: Radical Hysterectomy vs Simple Hysterectomy; Test type: Superiority; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.47 to 2.67] — Hazard ratio of simple to radical hysterectomy

3. Secondary Outcome: Extra-pelvic Relapse-free Survival
Description: It was defined as the time from randomization to the documented reappearance of disease provided that this recurrence is outside of pelvic. Patients who relapsed in pelvic field were censored at the time of first documented pelvic relapse. Patients who died before any relapse or alive without recurrence were censored at the date of death or last known alive date. 3 year extra-pelvic relapse-free survival was estimated by Kaplan-Meier method.
Time Frame: 3 years
Population: All patients randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radical Hysterectomy | Simple Hysterectomy
Number analyzed (Participants) | 350 | 350
percentage of participants | 99.7 [99.1 to 100.0] | 98.1 [96.6 to 99.6]
Statistical Analysis 1: Comparison: Radical Hysterectomy vs Simple Hysterectomy; Test type: Superiority; Hazard Ratio (HR) = 3.82, 95% CI 2-sided [0.79 to 18.4] — Hazard ratio is simple hysterectomy group of radical hysterectomy group

4. Secondary Outcome: Relapse-free Survival
Description: It was defined as the time from randomization to the first time when either a pelvic or extra-pelvic recurrence was documented. Patients who died before any recurrence or alive without recurrence were censored at the date of death or last known alive date. 3 year relapse-free survival was estimated by Kaplan-Meier method.
Time Frame: 3 years
Population: All patients randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radical Hysterectomy | Simple Hysterectomy
Number analyzed (Participants) | 350 | 350
percentage of participants | 97.8 [96.2 to 99.4] | 96.3 [94.2 to 98.4]
Statistical Analysis 1: Comparison: Radical Hysterectomy vs Simple Hysterectomy; Test type: Superiority; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.69 to 3.45] — Hazard ratio is simple hysterectomy group to radical hysterectomy group

5. Secondary Outcome: Overall Survival
Description: It was defined as the time from randomization until death from any cause. The living patients were censored at the date of last known alive. 3 year overall survival was estimated by Kaplan-Meier method.
Time Frame: 3 years
Population: All patients randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radical Hysterectomy | Simple Hysterectomy
Number analyzed (Participants) | 350 | 350
percentage of participants | 99.4 [98.5 to 100.0] | 99.1 [98.0 to 100.0]
Statistical Analysis 1: Comparison: Radical Hysterectomy vs Simple Hysterectomy; Test type: Superiority; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.38 to 3.14] — Hazard ratio of simple to radical hysterectomy

ADVERSE EVENTS:
Time Frame: Observed during the follow-up (up to 7 years after 4 weeks of surgery).
Description: Only adverse events related to surgery were collected from patients who had the surgery.
Arm/Group | Radical Hysterectomy | Simple Hysterectomy
All-Cause Mortality (participants affected / at risk) | 7/344 | 7/338
Serious Adverse Events (participants affected / at risk) | 0/344 | 0/338
Other Adverse Events (participants affected / at risk) | 208/344 | 181/338
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radical Hysterectomy (N=344) | Simple Hysterectomy (N=338)
Abdominal pain (Gastrointestinal disorders) | 47 | 36
Constipation (Gastrointestinal disorders) | 19 | 13
Fatigue (General disorders) | 28 | 19
Paresthesia (Nervous system disorders) | 22 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 13 | 21
Urinary incontinence (Renal and urinary disorders) | 38 | 16
Urinary retention (Renal and urinary disorders) | 34 | 2
Dyspareunia (Reproductive system and breast disorders) | 19 | 21
Pelvic pain (Reproductive system and breast disorders) | 17 | 23
Lymphedema (Vascular disorders) | 36 | 35
Hot flashes (Vascular disorders) | 20 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT01658930/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT01658930/SAP_001.pdf